CLINICAL TRIAL: NCT02926014
Title: Lingual Tonsil Hypertrophy Grading and Its Relation to Sociodemographic Factors and Clinical Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Klaipėda University (Other)
Responsible Party: Principal Investigator, Nora Siupsinskiene, Professor medical doctor of otorhinolaryngology, Lithuanian University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LTH1
Record Dates: First submitted 2016-08-27; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Lingual Tonsil Hypertrophy; Dysphagia
Keywords: Dysphagia; Lingual Tonsil Hypertrophy; Lingual Tonsil Enlargement
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lingual Tonsil Hypertrophy participants (Experimental): The research group consisted of 50 consecutive adult outpatients suffering from swallowing disorders, examined by otorhinolaryngologist at the Hospital of Lithuanian University of Health Sciences.
  Lingual Tonsil Hypertrophy was diagnosed using videolaryngoscopy.
  Interventions: Device: Videolaryngoscopy; Other: Reflux Symptom Index Questionnaire; Other: Dysphagia Screening Questionnaire
- Control participants (Other): The control group consisted of 50 healthy adult participants, who were examined using videolaryngoscopy and no pharyngeal pathologies were diagnosed, including lingual tonsil hypertrophy.
  Interventions: Device: Videolaryngoscopy; Other: Reflux Symptom Index Questionnaire; Other: Dysphagia Screening Questionnaire

INTERVENTIONS:
Device: Videolaryngoscopy — A rigid 70 degree laryngoscope is inserted into the subject's oropharynx, which allows to visualize the lingual tonsils. The size of the lingual tonsils is evaluated using DelGaudio and Friedman grading systems.
Other: Reflux Symptom Index Questionnaire — A validated clinical tool for suspecting laryngopharyngeal reflux (LPR). The questionnaire was proposed by Belafsky et al. (2002) and consists of 9 most common gastroesophageal reflux disease (GERD) and LPR symptoms: hoarseness or a problem with your voice; clearing your throat; excess throat mucus or postnasal drip; difficulty swallowing food, liquids, or pills; coughing after you ate or after lying down; breathing difficulties or choking episodes; troublesome or annoying cough; sensation of something sticking in your throat or a lump in your throat; heartburn, chest pain, indigestion, or stomach acid coming up. Each symptom is evaluated on a scale from 0 to 5 (0 - no complaint, 5 - severe symptom). The sum of all symptom evaluations ranges from 0 to 45.
Other: Dysphagia Screening Questionnaire — A validated questionnaire, proposed by Ohkuma et al. (2002). Lithuanian version of the questionnaire consists of 16 questions: choking during swallowing meals / liquids; difficulty eating solid foods; difficult swallowing; feeling of food getting stuck in the throat; longer than before eating time; feeling of food remaining in the mouth; feeling that food or liquid is going up into the throat from the stomach; feeling of food being stuck in the esophagus; weight loss; food getting stuck in the throat; food falling from the mouth; difficulty coughing during or after meals; occurrence of pneumonia; hoarseness; coughing during the night. Interpretation of dysphagia screening questionnaire:
  Advanced symptom - 2 points; Moderate intensity symptom - 1 point; No symptom - 0 point. At least one advanced symptom means - dysphagia. Higher score represents stronger dysphagia intensity. The maximum score is 32 points.

SUMMARY:
The aim of this research was to evaluate the lingual tonsil hypertrophy (LTH) grading of patients with dysphagia using videolaryngoscopy and determine the relation of LTH grades to sociodemographic factors and clinical symptoms.

DETAILED DESCRIPTION:
Two groups of people were interviewed during this research - the LTH group and the control group - a total of 100 subjects. The first group was comprised of 50 individuals, who visited the otorhinolaryngologist at Lithuanian University of Health Sciences hospital, regarding dysphagia, and were diagnosed with LTH during endoscopy. The second group consisted of 50 healthy individuals without dysphagia, who did not have enlarged lingual tonsils during assessment using videolaryngoscopy. All subjects filled out the questionnaires, composed of RSI (Reflux Symptom Index) and DSQ (Dysphagia Screening Questionnaire) questionnaires, validated and verified for use in Lithuania, together with a questionnaire created specifically for this research for gathering sociodemographic data.

The LTH grade of all subjects was determined using DelGaudio and Friedman grading systems.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Consent for participating in the research
* No cognitive disorders or mental illnesses
* Complaining about difficulty swallowing (research group)
* Enlarged lingual tonsils on videolaryngoscopy (research group)
* Generally healthy, no complaints of swallowing disorders (control group)
* Normal-sized lingual tonsils (control group)

Exclusion Criteria:

* Refusal to participate in the research
* Younger than 18 and older than 80 years old
* Serious mental or cognitive conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lingual tonsil enlargement grade on videolaryngoscopy | At baseline
  Lingual tonsil enlargement grade was assessed using DelGaudio (2008) and Friedman (2015) grading systems during videolaryngoscopy.
  According DelGaudio severity of LTH was assessed as: grade 0- lingual tonsils are not enlarged; 1- the lingual tonsils are prominent but not in full contact with the epiglottis or obscuring the valleculae; 2- the lingual tonsils obscure the view of the valleculae and are fully in contact with the epiglottis; 3- the lingual tonsils fill the valleculae and partially or fully obscure the view of the epiglottis.
  Friedman grading system consists of 0 to 4 scale: 0- complete absence of lymphoid tissue; 1- lymphoid tissue scattered over tongue base; 2- lymphoid tissue covering entirety of tongue base with limited vertical thickness; 3- significantly raised lymphoid tissue covering entirety of the tongue base, approximately 5 to 10 mm in thickness; 4- lymphoid tissue rising above the tip of the epiglottis, 10 or more mm in thickness.

SECONDARY OUTCOMES:
Sociodemographic factors: age | At baseline
  Participant's age in years at the time of the study.
Sociodemographic factors: gender | At baseline
  Gender: male/female.
Sociodemographic factors: body mass index (BMI) | At baseline
  Self-reported height and weight were used to calculate BMI (kg/m^2). Obesity was defined as a BMI value of 30 or higher, overweight as 25.0-29.9, normal weight as 18.5-24.9, and underweight as less than 18.5
Sociodemographic factors: occupation and employment status | At baseline
  Participants were asked about their job (job title). Occupations were classified as one of 4 categories: office worker; laborer; retired; disabled
Sociodemographic factors: health behaviors | At baseline
  Cigarette smoking status was categorised into 4 categories: "non smoker"; "smoker"; "former smoker"; "passive smoker". Lifetime alcohol drinking status was categorized according to the frequency of alcohol use as "never"; "several times a year"; "several times a month"; "several times a week".
Sociodemographic factors: previous tonsillectomy | At baseline
  Participants were asked if they had their palatal tonsils removed. if yes, they were asked how long ago it happened.
Sociodemographic factors: gastrointestinal diseases | At baseline
  The presence of gastrointestinal tract diseases was evaluated by asking participants if they were diagnosed with any disease of gastrointestinal tract. Most common were gastroesophageal reflux disease (GERD) and gastric/duodenal ulcers.
Sociodemographic factors: history of fibroesophagogastroduodenoscopy (FEGDS) findings | At baseline
  Data, found on FEGDS: erosive esophagitis (yes/no); hiatal hernia (yes/no); other gastric or duodenal pathologies.
Sociodemographic factors: use of antacids | At baseline
  We asked participants if they use antacid drugs, what kind of drug they use and the length of the use.
Sociodemographic factors: allergic diseases | At baseline
  History of allergic diseases: participants checked "yes" if they were diagnosed with an allergic disease; "no" if not.
General health status | At baseline
  General health status was selfreported using visual analogue scale (0-excellent/ very good, 10-poor).
Reflux Symptom Index questionnaire | At baseline
  A validated clinical tool for suspecting laryngopharyngeal reflux (LPR). The questionnaire consists of 9 most common gastroesophageal reflux disease (GERD) and LPR symptoms: hoarseness or a problem with your voice; clearing your throat; excess throat mucus or postnasal drip; difficulty swallowing food, liquids, or pills; coughing after you ate or after lying down; breathing difficulties or choking episodes; troublesome or annoying cough; sensation of something sticking in your throat or a lump in your throat; heartburn, chest pain, indigestion, or stomach acid coming up. Each symptom is evaluated on a scale from 0 to 5 (0 - no complaint, 5 - severe symptom). The sum of all symptom evaluations ranges from 0 to 45.
Dysphagia Screening Questionnaire | At baseline
  Lithuanian version of the questionnaire consists of 16 questions: choking during swallowing meals / liquids; difficulty eating solid foods; difficult swallowing; feeling of food getting stuck in the throat; longer than before eating time; feeling of food remaining in the mouth; feeling that food or liquid is going up into the throat from the stomach; feeling of food being stuck in the esophagus; weight loss; food getting stuck in the throat; food falling from the mouth; difficulty coughing during or after meals; occurrence of pneumonia; hoarseness; coughing during the night. Interpretation of dysphagia screening questionnaire:
  Advanced symptom - 2 points; Moderate intensity symptom - 1 point; No symptom - 0 point. At least one advanced symptom means - dysphagia. Higher score represents stronger dysphagia intensity. The maximum score is 32 points.
Symptom severity | At baseline
  Participants were asked to evaluate 8 most common LTH symptoms using visual analogue scale (10 cm line, where 0 cm- no symptom, 10 cm- extremely severe symptom). Symptoms: hoarseness; difficult swallowing; painful swallowing; sensation of something sticking in your throat or a lump in your throat; difficult breathing, shortness of breath; snoring; cough; pain in the neck, pharynx.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Siupsinskiene, Professor, Principal Investigator — Hospital of Lithuanian University of Health Sciences, Otorhinolaryngology department; Nora Siupsinskiene, Professor, Principal Investigator — Klaipėda University
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania